CLINICAL TRIAL: NCT06551194
Title: Prevalence, Characteristics, Management, and Outcomes of Difficult-to-treat Inflammatory Bowel Disease: Multicenter Retrospective Study
Brief Title: Prevalence, Characteristics, Management, and Outcomes of Difficult-to-treat Inflammatory Bowel Disease
Acronym: DTT-IBD
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Tommaso Lorenzo Parigi, MD Gastroenterologist, IRCCS Ospedale San Raffaele
Other Study IDs: DTT-IBD
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Assessment of the Criteria and Risk Factors for DTT-IBD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UC patients: Adult patients (age ≥18) diagnosed with UC
  Interventions: Other: prevalence of difficult-to-treat IBD
- CD patients: Adult patients (age ≥18) diagnosed with UC
  Interventions: Other: prevalence of difficult-to-treat IBD

INTERVENTIONS:
Other: prevalence of difficult-to-treat IBD — To assess the prevalence and risk factors of difficult-to-treat IBD patients

SUMMARY:
Crohn's disease (CD) and ulcerative colitis (UC) are the two main types of chronic inflammatory bowel disease (IBD). Despite recent advances, many patients do not respond to available treatments and or lose response over time.

In 2023, the International Organisation for the Study of IBD (IOIBD) proposed a common definition of 'difficult-to-treat' inflammatory bowel disease (IBD-IBD) to homogenise terminology and promote research into patients most in need of new treatments and therapeutic strategies. According to the IOIBD criteria, IBD is defined by any of the following: failure of two or more advanced treatments with different mechanisms of action, postoperative recurrence of Crohn's disease after two or more bowel resections, pouchitis refractory to antibiotics, complex perianal Crohn's disease, or the presence of psychiatric comorbidity that prevents adequate therapeutic management.

As the definition of DTT-IBD is very recent, the prevalence and risk factors of DTT-IBD are not yet known. This study aims to determine the prevalence of DTT-IBD in the patient population and the risk factors associated with the development of DTT-IBD. The study will be conducted as a retrospective cross-sectional study in two large tertiary care centers, IRCCS Ospedale San Raffaele and IRCCS Humanitas Research Hospital, both in Milan, Italy. The study will evaluate the criteria and risk factors for DTT-IBD in the latest available gastroenterological examination report, provided it was performed in the last 5 years (from 1 January 2019).

DETAILED DESCRIPTION:
This is a multicentre retrospective cross-sectional study with two aims:

1. To evaluate the prevalence of difficult-to-treat IBD
2. To evaluate which and how demographic and clinical variables affect the risk of DTT-IBD

The subjects considered are adult patients (≥18 years) diagnosed with UC or CD followed at San Raffaele Hospital and Humanitas Research Hospital.

Crohn's disease (CD) and ulcerative colitis (UC) are the two main types of chronic inflammatory bowel disease (IBD). Despite recent advances, many patients do not respond to available treatments and or lose response over time.

In 2023, the International Organisation for the Study of IBD (IOIBD) proposed a common definition of 'difficult-to-treat' inflammatory bowel disease (IBD-IBD) to homogenise terminology and promote research into patients most in need of new treatments and therapeutic strategies. According to the IOIBD criteria, IBD is defined by any of the following: failure of two or more advanced treatments with different mechanisms of action, postoperative recurrence of Crohn's disease after two or more bowel resections, pouchitis refractory to antibiotics, complex perianal Crohn's disease, or the presence of psychiatric comorbidity that prevents adequate therapeutic management.

As the definition of DTT-IBD is very recent, the prevalence and risk factors of DTT-IBD are not yet known. This study aims to determine the prevalence of DTT-IBD in the patient population and the risk factors associated with the development of DTT-IBD. The study will be conducted as a retrospective cross-sectional study in two large tertiary care centers, IRCCS Ospedale San Raffaele and IRCCS Humanitas Research Hospital, both in Milan, Italy. The study will evaluate the criteria and risk factors for DTT-IBD in the latest available gastroenterological examination report, provided it was performed in the last 5 years (from 1 January 2019).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18)
* Diagnosis of IBD: Crohn's disease (CD), ulcerative colitis (UC), or undetermined IBD (IBD-U)
* A least one visit with a gastroenterology specialist after 01/01/2019

Exclusion Criteria:

* Unconfirmed IBD diagnosis
* Consultation with non-gastroenterology specialists
* Consultation older than January 1st 2019
* Pediatric patients (Age <18). Pediatric population will be excluded as the DTT-IBD criteria apply to adult patients only.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18) diagnosed with IBD followed at San Raffaele Hospital and Humanitas Hospital
Sampling Method: Probability Sample
Enrollment: 972 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
IBD not meeting the DTT-IBD criteria | 3 months
  In absence of prior literature describing the prevalence of DTT (our will be the first study) a sample size calculation can only be estimated based on clinical experience.
  Based on our clinical experience, assuming a Cohen effect size of 0.18, using a two-sided t-test with an alfa error of 0.05, 486 subjects in each group would be needed to detect a significant difference between the two (DTT and non-DTT). Therefore the total included population would be 486 x 2 = 972 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Lo Parigi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy